CLINICAL TRIAL: NCT03776240
Title: A Phase I, Double-Blind, Randomised, Parallel Group Study to Demonstrate the Equivalent Pharmacokinetic Properties of a Single Intravenous Dose of HD201 and EU-Herceptin® and US-Herceptin® in Healthy Male Subjects
Brief Title: A Study to Demonstrate the Equivalent Pharmacokinetic Properties of a Single Intravenous Dose of HD201 and EU-Herceptin® and US-Herceptin® in Healthy Male Subjects
Acronym: TROIKA-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Prestige Biopharma Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: TROIKA-1
Record Dates: First submitted 2018-12-13; First posted 2018-12-14 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2023-02

CONDITIONS: Healthy Volunteers
Keywords: randomized; double-blind
MeSH Terms: interventions — Trastuzumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- HD201 (Experimental): Trastuzumab Single-dose 6mg/kg body weight by 90 minute intravenous infusion
  Interventions: Drug: HD201
- EU-licensed Herceptin (Active Comparator): Trastuzumab Single-dose 6mg/kg body weight by 90 minute intravenous infusion
  Interventions: Drug: EU-Herceptin
- US-licensed Herceptin (Active Comparator): Trastuzumab Single-dose 6mg/kg body weight by 90 minute intravenous infusion
  Interventions: Drug: US-Herceptin

INTERVENTIONS:
Drug: HD201 — Single-dose 6mg/kg body weight by 90 minute intravenous infusion
  Other Names: Trastuzumab
  Arms: HD201
Drug: EU-Herceptin — Single-dose 6mg/kg body weight by 90 minute intravenous infusion
  Other Names: Trastuzumab
  Arms: EU-licensed Herceptin
Drug: US-Herceptin — Single-dose 6mg/kg body weight by 90 minute intravenous infusion
  Other Names: Trastuzumab
  Arms: US-licensed Herceptin

SUMMARY:
The purpose of the study is to demonstrate demonstrate the pharmacokinetic (PK) similarity of HD201 to the European (EU) and American (US) reference products Herceptin, following a single i.v. infusion of 6 mg/kg in healthy volunteers.

DETAILED DESCRIPTION:
This is a double-blind, randomised, parallel group study, where a total of 105 healthy adult male volunteers, ≥ 18 and ≤ 55 years of age, non-smoker, will be dosed; 35 subjects per treatment group, randomly assigned to one of the 3 treatment arms.

ELIGIBILITY:
Inclusion Criteria:

1. Male, non-smoker (no use of tobacco products within 3 months prior to screening), ≥ 18 and ≤ 55 years of age, with BMI > 18.5 and < 30.0 kg/m2 and body weight ≥ 50.0 kg.
2. Healthy as defined by:

   1. the absence of clinically significant illness and surgery within 4 weeks prior to dosing. Inclusion pre-dosing is at the discretion of the Principal Investigator.
   2. the absence of clinically significant history of neurological, endocrinal, cardiovascular, pulmonary, hematological, immunologic, psychiatric, gastrointestinal, renal, hepatic, and metabolic disease.
   3. a LVEF within the normal range as measured by echocardiogram (ECHO) within 4 weeks prior to randomization.
   4. the absence of clinically significant history of anaphylaxis, angioedema, interstitial pneumonitis, or acute respiratory distress syndrome.
3. Male subjects who are not vasectomized for at least 6 months, and who are sexually active with non-sterile female partner [sterile female partners include post-menopausal women (absence of menses for 12 months prior to drug administration) or women who have had a tubal ligation, hysterectomy, or bilateral oophorectomy (at least 6 months prior to drug administration)] must be willing to use one of the following acceptable contraceptive method throughout the study and for 90 days after the last study drug administration:

   1. simultaneous use of condom, and for the female partner hormonal contraceptives (used since at least 4 weeks) or intra-uterine contraceptive device (placed since at least 4 weeks);
   2. simultaneous use of male condom, and for the female partner, diaphragm with intravaginally applied spermicide.
4. Male subjects, including men who have had vasectomy, with a pregnant partner must agree to use a condom throughout the study and for 90 days after the last study drug administration.
5. Male subjects must be willing not to donate sperm until 90 days following the last study drug administration.
6. Capable of consent.

Exclusion Criteria:

f the following applies will be excluded from the study:

1. Any clinically significant abnormality or abnormal laboratory test results found during medical screening or positive test for hepatitis B, hepatitis C, or HIV found during medical screening.
2. Positive urine drug screen at screening.
3. History of allergic reactions to trastuzumab, benzyl alcohol, murine proteins, or other related drugs.
4. Any reason which, in the opinion of the Principal Investigator, would prevent the subject from participating in the study.
5. Clinically significant ECG abnormalities (QTc >450 ms) and or vital sign abnormalities (systolic blood pressure lower than 90 or over 140 mmHg, diastolic blood pressure lower than 50 or over 90 mmHg, or heart rate less than 50 or over 100 bpm) at screening.
6. History of significant alcohol abuse within one year prior to screening or regular use of alcohol within six months prior to the screening visit (more than fourteen units of alcohol per week [1 unit = 150 mL of wine, 360 mL of beer, or 45 mL of 40% alcohol]).
7. History of significant drug abuse within one year prior to screening or use of soft drugs (such as marijuana) within 3 months prior to the screening visit or hard drugs (such as cocaine, phencyclidine [PCP], crack, opioid derivatives including heroin, and amphetamine derivatives) within 1 year prior to screening.
8. Previous use of trastuzumab or another monoclonal antibody for a medical condition or in the context of another clinical trial.
9. Participation in a clinical research study involving the administration of an investigational or marketed drug or device within 30 days prior to the first dosing, administration of a biological product in the context of a clinical research study within 90 days prior to the first dosing, or concomitant participation in an investigational study involving no drug or device administration.
10. Use of medication other than topical products without significant systemic absorption:

    1. prescription medication within 14 days prior to dose administration;
    2. over-the-counter products including natural health products (e.g. food supplements and herbal supplements) within 7 days prior to dosing, with the exception of the occasional use of acetaminophen (paracetamol - up to 2 g daily);
    3. a depot injection or an implant of any drug within 3 months prior to dose administration.
11. Donation of plasma within 7 days prior to dosing. Donation or loss of blood (excluding volume drawn at screening) of 50 mL to 499 mL of blood within 30 days, or more than 499 mL within 56 days prior to the first dosing.
12. Hemoglobin < 12.8 g/dL and hematocrit < 0.37 L/L at screening.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-08-19 (Actual); Study Completion 2019-08-19 (Actual)

PRIMARY OUTCOMES:
Area under Curve (AUC, Pharmacokinetics) | Up to day 54
  Sampling will be performed in all patients to compare PK though values of HD201 and Herceptin

SECONDARY OUTCOMES:
Immunogenicity: Incidence of anti-herceptin antibodies | 0 hour, Day 15, Day 29, Day 43, and Day 54 post-dose
  Incidence of anti-herceptin antibodies

CONTACTS AND LOCATIONS:
Locations (1):
- Q Pharm, Brisbane, Australia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Demarchi M, Coliat P, Mclendon K, Chung Shii Hii J, Feyaerts P, Ang F, Jaison L, Deforce F, Derde MP, Kim MJ, Park LS, Detappe A, Pivot X. TROIKA-1: A double-blind, randomized, parallel group, study aimed to demonstrate the equivalent pharmacokinetic profile of HD201, a potential biosimilar candidate to trastuzumab, versus EU-Herceptin(R) and US-Herceptin(R) in healthy male subjects. Pharmacol Res Perspect. 2021 Aug;9(4):e00839. doi: 10.1002/prp2.839. PMID 34309241